CLINICAL TRIAL: NCT03216070
Title: Low-dose Dasatinib as First-line Treatment for Chronic Myeloid Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dra. Olga Graciela Cantu Rodriguez, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE17 00004
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Dasatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm1 Low Dose Dasatinib (Experimental): We will give 50mg of dasatinib orally daily for 6 months
  Interventions: Drug: Dasatinib 50 MG

INTERVENTIONS:
Drug: Dasatinib 50 MG — 50mg of dasatinib orally daily
  Other Names: Sprycel

SUMMARY:
Our goal is to demonstrate that 50mg of dasatinib is as effective as the full dose to induce molecular response as first line therapy in CML.

DETAILED DESCRIPTION:
We will give 50mg of dasatinib daily since the diagnosis for up to 6 months, for the first 2-4 weeks we will evaluate hematic biometry to registry hematic response, at months 3 and 6 a BCR/ABL PCR will be taken to evaluate molecular response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BCR-ABL positive CML in early chronic phase CML. Except for hydroxyurea, patients must have received no or minimal prior therapy, defined as <2 weeks (14 days) of prior FDA approved TKI.
* ECOG performance of 0-2
* Adequate end organ function, defined as the following: total bilirubin <1.5x ULN, SGPT <2.5x ULN, creatinine <1.5x ULN.
* Patients must sign an informed consent indicating they are aware of the investigational nature of this study.

Exclusion Criteria:

* NYHA cardiac class 3-4 heart disease or previous pleural effusion.
* Pregnancy and lactation
* Patients with active, uncontrolled psychiatric disorders

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Molecular Response at 6 months | 6 months
  Molecular Response define as BCR/ABL <1%

SECONDARY OUTCOMES:
Early Molecular Response at 3 and 6 months | 3 and 6 months
  Early Molecular Response define as <10%

CONTACTS AND LOCATIONS:
Locations (1):
- Hopsital Universitario Dr. Jose E. Gonzalez, Centro Universitario contra el Cancer, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keskin D, Sadri S, Eskazan AE. Dasatinib for the treatment of chronic myeloid leukemia: patient selection and special considerations. Drug Des Devel Ther. 2016 Oct 13;10:3355-3361. doi: 10.2147/DDDT.S85050. eCollection 2016. PMID 27784993
- [Background] Stein B, Smith BD. Treatment options for patients with chronic myeloid leukemia who are resistant to or unable to tolerate imatinib. Clin Ther. 2010 May;32(5):804-20. doi: 10.1016/j.clinthera.2010.05.003. PMID 20685492
- [Background] Tokarski JS, Newitt JA, Chang CY, Cheng JD, Wittekind M, Kiefer SE, Kish K, Lee FY, Borzillerri R, Lombardo LJ, Xie D, Zhang Y, Klei HE. The structure of Dasatinib (BMS-354825) bound to activated ABL kinase domain elucidates its inhibitory activity against imatinib-resistant ABL mutants. Cancer Res. 2006 Jun 1;66(11):5790-7. doi: 10.1158/0008-5472.CAN-05-4187. PMID 16740718
- [Background] Kantarjian H, Shah NP, Hochhaus A, Cortes J, Shah S, Ayala M, Moiraghi B, Shen Z, Mayer J, Pasquini R, Nakamae H, Huguet F, Boque C, Chuah C, Bleickardt E, Bradley-Garelik MB, Zhu C, Szatrowski T, Shapiro D, Baccarani M. Dasatinib versus imatinib in newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2010 Jun 17;362(24):2260-70. doi: 10.1056/NEJMoa1002315. Epub 2010 Jun 5. PMID 20525995
- [Background] Shah NP, Kantarjian HM, Kim DW, Rea D, Dorlhiac-Llacer PE, Milone JH, Vela-Ojeda J, Silver RT, Khoury HJ, Charbonnier A, Khoroshko N, Paquette RL, Deininger M, Collins RH, Otero I, Hughes T, Bleickardt E, Strauss L, Francis S, Hochhaus A. Intermittent target inhibition with dasatinib 100 mg once daily preserves efficacy and improves tolerability in imatinib-resistant and -intolerant chronic-phase chronic myeloid leukemia. J Clin Oncol. 2008 Jul 1;26(19):3204-12. doi: 10.1200/JCO.2007.14.9260. Epub 2008 Jun 9. PMID 18541900